CLINICAL TRIAL: NCT02478021
Title: Effekte Von Hydrocortison Auf Soziale Kognition Und Gedächtnis Unter Berücksichtigung Von Geschlechtereffekten
Brief Title: Effects of Hydrocortisone on Social Cognition and Memory
Acronym: CORT-COG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Katja Wingenfeld, PhD, Head: Clinical Psycology, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: WI-CO-1
Record Dates: First submitted 2015-06-11; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Individuality
Keywords: effects of cortisol on cognition
MeSH Terms: interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrocortisone (Experimental): 10 mg hydrocortisone
  Interventions: Other: Hydrocortisone
- Placebo (Placebo Comparator): 1 pill Placebo
  Interventions: Other: Hydrocortisone

INTERVENTIONS:
Other: Hydrocortisone — Effects of hydrocortisone compared to placebo on cognition

SUMMARY:
The effects of hydrocortisone on cognition will be investigated.

DETAILED DESCRIPTION:
80 healthy young individuals (40 females and 40 male) will be recruited an randomized to either placebo or 10 mg hydrocortisone before testing. Tasks will on emotion recognition, memory and cognitive flexibilty will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 30
* medication free

Exclusion Criteria:

* any medication
* severe ilness

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
social cognition | 25 min
  computer based test: Multifaceted Empaty test

SECONDARY OUTCOMES:
memory | 25 min
  autobiographic memory test (AMT)
cognitive flexibilty | 10 min
  computer based test: task switch

CONTACTS AND LOCATIONS:
Overall Officials: Katja Wingenfeld, Principal Investigator — Charite University
Locations (1):
- Charite University, Berlin, Germany